CLINICAL TRIAL: NCT03004222
Title: A Randomized Double Blinded Study to Determine the Effectiveness of Utilizing Intraperitoneal Bupivacaine: Does it Reduce Post-operative Opioid Use Following Laparoscopic Appendectomy?
Brief Title: A Study to Determine the Effectiveness of Utilizing Intraperitoneal Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metro Health, Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Appendectomy Study
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopic Appendectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anesthetic (Bupivicaine) (Experimental): The experimental arm intervention is 75 subjects will receive the study agent (20 mL of 0.5% bupivacaine) to be sprayed at the cecum after the appendix has been removed and all planned irrigation and aspiration has occurred
  Interventions: Drug: Bupivacaine
- Placebo 20 ml (Placebo Comparator): 75 subjects will be treated with normal saline/placebo to be sprayed at the cecum after the appendix has been removed and all planned irrigation and aspiration has occurred
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Bupivacaine — 20 ml of 0.5% Bupivacaine
  Arms: Local anesthetic (Bupivicaine)
Drug: Placebos
  Arms: Placebo 20 ml

SUMMARY:
The purpose of this research is to determine if spraying a local anesthetic to the cecum after a laparoscopic appendectomy decreases the amount of narcotics (pain medicine) needed after surgery and reduces the time to discharge from the hospital.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of using intraperitoneal anesthetic during appendectomy. Subjects will be randomized to receive either 20 mL 0.5% bupivicaine or 20 mL of normal saline (placebo) instilled in the right lower quadrant at the cecum after appendix has been removed. Narcotic consumption will be tracked postoperatively. Hypothesis is that instilling local anesthetic at the cecum during a laparoscopic appendectomy will decrease the amount of narcotic a patient uses postoperatively. Secondarily, this study will attempt to determine if there is a decrease in length of stay for the subjects randomized to the anesthetic infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Laparoscopic appendectomy at Metro Health Hospital

Exclusion Criteria:

* Adults unable to consent Non-English speaking patients
* Suspected or known malignant disease
* Patients with known allergies to the local anesthetic
* Utilizes opioid pain medicine for a chronic condition
* Elective laparoscopic appendectomy
* Known allergy or contraindication to ketorolac

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Total narcotic use following surgery until the time of discharge from the hospital. | 1, 2, 4 hours

SECONDARY OUTCOMES:
Time to Discharge | 12 hours
Pain Level Scores at 1, 2, 4, and 12 hours postoperatively | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karlin Sevensma, DO, Principal Investigator — Metro Health Hospital
Locations (1):
- Metro Health Hospital, Wyoming, Michigan, United States

IPD SHARING:
Plan to Share IPD: No